# **Informed Consent Form**

**TITLE:** Better Together: A Patient-centered Approach to Improve Diabetes Among Immigrant Communities

NCT NUMBER: NCT05275231

IRB APPROVAL DATE: November 12, 2021

# You Are Being Asked to Be in a Research Study

Concise presentation of key concepts

You are being asked to be in a research study. A research study is designed to answer a scientific question. If you agree to be in the study you will be one of 48 people who are being studied, at Emory.

# Why is this study being done?

This study is being done to answer the question: are culturally tailored group visits feasible and acceptable among South Asian immigrant populations with diabetes or prediabetes. You are being asked to be in this research study because you meet our study criteria and may benefit from this study.

# Do you have to be in the study?

It is your decision to be part of this research study. You do not have to be in it. Your choice will not affect your access to medical care for your condition. Before you make your decision, you should take time to learn about the study.

# What do I have to do if I choose to participate in this study?

If you are eligible and want to be part of the study, you will participate for 5 months(5 in group virtual sessions over 16 weeks). The researchers will ask you to do the following: complete a paper survey, get a health assessment including weight, blood pressure reading, and A1c check by a droplet of blood. All of these procedures will be paid for by the study.

# How is this study going to help you?

If you are in the study, you will be helping the researchers answer the study question. This study is designed to benefit you directly. You will be provided with free education materials and guidance on health lifestyle choices to manage your health. In addition, the study results may be used to help others in the future.

# What are the risks or discomforts I should know about before making a decision?

The study will take time. All studies have some risks. Some risks are relatively small, like being bored or losing time. Some are more serious – for this study, these include, loss of privacy, and breach of confidentiality. A full list of expected risks, their frequency and severity are in the "What are the possible risks and discomforts?" section of this document.

Version Date: 10/25/2021



# **Alternatives to Joining This Study**

The alternatives include not joining the study and continuing to receive your usual care from y our primary care provider.

## Costs

You WILL NOT have to pay for any of the study procedures, in particular those that are not covered by your medical insurance.

## What Should I Do Next?

Read this form, or have it read to you. Make sure the study doctor or study staff explains the study to you. Ask questions (e.g., about exact time commitment, about unfamiliar words, more details on specific procedures, etc.) Take time to consider this, and talk about it with your family and friends.

\*\*A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

 Version Date: 10/25/2021



# Emory University Consent to be a Research Subject

<u>Title</u>: Better Together: A patient-centered approach to improve diabetes among immigrant communities

<u>Principal Investigator:</u> Megha K. Shah, MD, MSc; Department of Family and Preventive Medicine, Emory School of Medicine

## **Funding Source:**

National Institute on Minority Health and Health Disparities

#### Introduction

You are being asked to be in a research study. This form is designed to tell you everything you need to think about before you decide to consent (agree) to be in the study or not to be in the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. You can skip any questions that you do not wish to answer.

Before making your decision:

- Please carefully read this form or have it read to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. By signing this form you will not give up any legal rights.

#### **Study Overview**

The purpose of this study is to determine if a tailored lifestyle intervention is acceptable and feasible for South Asian immigrants with diabetes or prediabetes.

#### **Procedures**

Your participation is voluntary. You will be asked to participate in a 16-week lifestyle program. There will be a total of 5 virtual group sessions. You will be provided with health education materials and guidance on how to improve your diet to reduce your risk of diabetes or improve your diabetes management. Each session will last about 60-90 minutes. While we encourage you to participate in all the sessions, your participation is voluntary.

Over the course of your participation, we will collect some basic health information. This will include your height, weight, blood pressure, and finger prick testing of glucose and cholesterol. The finger prick testing will occur at the beginning and end of the study, and 1 year after the study ends.

#### Who owns my study information and samples?

If you join this study, you will be donating your study information. You will not receive any compensation if your samples or information are used to make a new product

#### **Risks and Discomforts**

The most common risks and discomforts expected in this study are: anxiety related to participating in group visits. We will collect samples via finger prick testing at the beginning and end of the study, there may be some minor pain associated with this, and a very low risk of infection. Measures will be taken to keep this risk minimal. There is a risk of

Version Date: 10/25/2021

 IRB Form 01242020



loss of confidentiality of study data. We will, however, take measures to ensure that this does not happen. No other risks are known.

#### Will I benefit directly from the study?

Your diabetes/prediabetes may improve while you are in this study but it may not, and it may even get worse. This study is designed to learn more about preferences for diabetes related health education. The study results may be used to help others in the future.

#### Will I be compensated for my time and effort?

You will get a \$20 gift card for each completed study survey, to compensate you for your time and effort. If you do not finish the study, we will compensate you for the surveys you have completed. You will get \$75 total in gift cards, if you complete all study visits. You may be asked to fill out a tax form, including your Social Security or Taxpayer Identification Number, in order to be reimbursed, depending on the amount and method of payment. Some payment methods involve mail coming to your house, which may be seen by others in your household. You can decline payment if you are concerned about confidentiality, or you can talk to the study team to see if there are other payment options.

#### **New Information**

It is possible that the researchers will learn something new during the study about the risks of being in it. If this happens, they will tell you about it. Then you can decide if you want to continue to be in this study or not. You may be asked to sign a new consent form that includes the new information if you decide to stay in the study.

#### **Benefits**

This study is designed to benefit you directly. You will be provided with free education materials and guidance on health lifestyle choices to manage your health. In addition, the study results may be used to help others in the future.

#### Compensation

You will get a \$20 gift card for each data collection timepoint. You will receive an additional \$35 for completing the education sessions. If you do not finish the study, you will be paid for the visits and sessions that you have completed. You will receive \$75 total in gift cards if you complete all study visits. Some payment methods involve mail coming to your house, which may be seen by others in your household. You can decline payment if you are concerned about confidentiality, or you can talk to the study team to see if there are other payment options.

#### **Other Options Outside this Study**

If you decide not to enter this study, there is care available to you outside of this research. You can still receive routine care from your primary care provider. We will discuss these with you. You do not have to be in this study to be treated for diabetes/prediabetes

#### How will you protect my private information that you collect in this study?

Whenever possible, a study number, rather than your name, will be used on study records. Your name and other identifying information will not appear when we present or publish the study results.

Certain offices and people other than the researchers may look at study records. Government agencies and Emory employees overseeing proper study conduct may look at your study records. These offices include the Office for Human Research Protections, the funder(s), the Emory Institutional Review Board, the Emory Office of Research Compliance.

 Version Date: 10/25/2021

IRB Form 01242020



Study funders may also look at your study records. Emory will keep any research records we create private to the extent we are required to do so by law. A study number rather than your name will be used on study records wherever possible. Your name and other facts that might point to you will not appear when we present this study or publish its results.

#### **Certificate of Confidentiality**

There is a Certificate of Confidentiality from the National Institutes of Health for this Study. The Certificate of Confidentiality helps us to keep others from learning that you participated in this study. Emory will rely on the Certificate of Confidentiality to refuse to give out study information that identifies you. For example, if Emory received a subpoena for study records, it would not give out information that identifies you.

The Certificate of Confidentiality does not stop you or someone else, like a member of your family, from giving out information about your participation in this study. For example, if you let your insurance company know that you are in this study, and you agree to give the insurance company research information, then the investigator cannot use the Certificate to withhold this information. This means you and your family also need to protect your own privacy.

The Certificate does not stop Emory from making the following disclosures about you:

- Giving state public health officials information about certain infectious diseases,
- Giving law officials information about abuse of a child, elderly person or disabled person.
- Giving out information to prevent harm to you or others.

Giving the study sponsor or funders information about the study, including information for an audit or evaluation.

#### **Storing and Sharing your Information**

De-identified data from this study (data that has been stripped of all information that can identify you), may be placed into public databases where, in addition to having no direct identifiers, researchers will need to sign data use agreements before accessing the data. We will remove or code any personal information that could identify you before your information is shared. This will ensure that, by current scientific standards and known methods, it is extremely unlikely that anyone would be able to identify you from the information we share. Despite these measures, we cannot guarantee anonymity of your personal data.

Your data from this study may be useful for other research being done by investigators at Emory or elsewhere. To help further science, we may provide your deidentified data to other researchers. If we do, we will not include any information that could identify you. If your data or specimens are labeled with your study ID, we will not allow the other investigators to link that ID to your identifiable information.

We will use your sample and data only for research. We will not sell them.

As they become available, do you want us to contact you and ask whether you want to receive your results? If so, let the study team know, and they will contact you as the results become available.

#### Costs

There will be no costs to you for participating in this study, other than basic expenses like transportation. You will not be charged for any of the research activities.

 Version Date: 10/25/2021 IRB Form 01242020



#### Withdrawal from the Study

You have the right to leave a study at any time without penalty.

The researchers also have the right to stop your participation in this study without your consent for any reason, especially if they believe it is in your best interest or if you were to object to any future changes that may be made in the study plan.

These are the expected reasons why the researchers may stop your participation:

• If you experience any life-threatening condition or condition that prevents you from participating in moderate physical activity.

# **Authorization to Use and Disclose Protected Health Information**

The privacy of your health information is important to us. As part of this study, we will be requesting health care entities who are covered by the Health Insurance Portability and Accountability Act and regulations (HIPAA) to provide us with health information that identifies you ("individually identifiable health information" or "IIHI"). Because the health care entities are covered by HIPAA, we must have your authorization to obtain your IIHI from them. However, the researchers who get your IIHI from the health care entities are not covered by HIPAA. Once they receive your IIHI from the health care entities, they will put it in a separate research record that is not a part of your medical record. IIHI placed in the separate research record is not be covered by HIPAA.

#### **Purpose of this Authorization:**

By signing this form, you give us permission to get your IIHI from health care entities and to use and share your IIHI as described in this document. You do not have to sign this form. If you do not sign this form, then you may not participate in the research study.

#### **Research-Related Treatment**

This study involved research-related treatment that will not be electronically billed to any insurance company or government benefits program (e.g., Medicare, Medicaid). You may not receive the research-related treatment unless you sign this authorization. You may receive any non-research related treatment whether or not you sign this form.

## IIHI that Will be Used/Disclosed:

The IIHI that we will use or share for the research study includes:

- Medical information about you including your medical history and present/past medications.
- Laboratory test results.

## Purposes for Which Your IIHI Will be Used/Disclosed:

We will use and share your IIHI for the conduct and oversight of the research study. Once we have your IIHI we will keep it in a separate research record that will be used for the conduct of the study. If you leave the study, we may use your IIHI to determine your vital status or contact information.

#### People Who will Use/Disclose Your IIHI:

The following people and groups will use and disclose your IIHI in connection with the research study:

• The Principal Investigator and the research staff will use and disclose your IIHI to conduct the study.

Version Date: 10/25/2021

 IRB Form 01242020

- The Principal Investigator and research staff will share your IIHI with other people and groups to help conduct the study or to provide oversight for the study. This includes sharing your IIHI with people and groups at other sites who are helping conduct the study.
- NIMHD is the Sponsor of the study. The Sponsor may use and disclose your IIHI to make sure the
  research is done correctly and to collect and analyze the results of the research. The Sponsor may
  disclose your IIHI to other people and groups like study monitors to help conduct the study or to provide
  oversight for the study.
- The following people and groups will use your IIHI to make sure the research is done correctly and safely:
  - Emory offices that are part of the Human Research Participant Protection Program and those that are involved in study administration. These include the Emory IRB, the Emory University and Healthcare Compliance Offices, and the Emory Office for Clinical Research.
  - Government agencies that regulate the research including: Office for Human Research Protections.
  - o Public health agencies.
  - o Research monitors and reviewer.
  - Accreditation agencies.
- Sometimes a Principal Investigator or other researcher moves to a different institution. If this happens, your IIHI may be shared with that new institution and their oversight offices.

#### **Expiration of Your Authorization**

Your IIHI will be used until this research study ends.

# **Revoking Your Authorization**

If you sign this form, at any time later you may revoke (take back) your permission to use your IIHI. If you want to do this, you must contact the study team at:

At that point, the researchers would not collect any more of your IIHI. But they may use or disclose the information you already gave them as described in this Authorization. If you revoke your authorization you will not be able to stay in the study.

#### Other Items You Should Know about Your Privacy

Not all people and entities are covered by the Privacy Rules. HIPAA only applies to health care providers, health care payers, and health care clearinghouses. HIPAA does not apply to research that does not include treatment that is billed to insurers or government benefit programs. If we disclose your information to people who are not covered by the Privacy Rules, including HIPAA, then your information won't be protected by the Privacy Rules. People who do not have to follow the Privacy rules can use or disclose your information with others without your permission if they are allowed to do so by the laws that cover them. The researchers and people and companies working with them are not covered by the Privacy Rules. They will only use and disclose your information as described in this Consent and Authorization.

To maintain the integrity of this research study, you generally will not have access to your IIHI related to this research until the study is complete. When the study ends, and at your request, you generally will only have access to your IIHI that we maintain in a designated record set. A designated record set is data that includes medical information or billing records that your health care providers use to make decisions about you. You will not have a right of access to IIHI kept in a separate research record used only for research purposed. If it is necessary for your health care, your health information will be provided to your doctor.

Version Date: 10/25/2021

 IRB Form 01242020



We may remove identifying information from your IIHI. Information without identifiers is not subject to HIPAA and may be used or disclosed with other people or organizations for purposes besides this study.

## **Contact Information**

Contact

- if you have any questions about this study or your part in it,
- if you have questions, concerns or complaints about the research

Contact the Emory Institutional Review Board at 404-712-0720 or 877-503-9797 or irb@emory.edu:

- if you have questions about your rights as a research participant.
- if you have questions, concerns or complaints about the research.
- You may also let the IRB know about your experience as a research participant through our Research Participant Survey at <a href="http://www.surveymonkey.com/s/6ZDMW75">http://www.surveymonkey.com/s/6ZDMW75</a>.

# **Consent and Authorization**

| TO BE FILLED OUT BY SUBJECT Please print your name, sign, and date below if you agree to be in this reauthorization form, you will not give up any of your legal rights. | | gning this consent and |
|---|---|---|
| Name of Subject | _ | |
| Signature of Subject (18 or older and able to consent) | | Time |
| TO BE FILLED OUT BY STUDY TE | EAM ONLY | |
| Name of Person Conducting Informed Consent Discussion | | |
| Signature of Person Conducting Informed Consent Discussion | | Time |

 Version Date: 10/25/2021 IRB Form 01242020